CLINICAL TRIAL: NCT04770779
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Mitapivat in Subjects With Transfusion-Dependent Alpha- or Beta-Thalassemia (ENERGIZE-T)
Brief Title: A Study Evaluating the Efficacy and Safety of Mitapivat in Participants With Transfusion-Dependent Alpha- or Beta-Thalassemia (α- or β-TDT)
Acronym: ENERGIZE-T
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG348-C-018; 2021-000212-34 (EudraCT Number); 2024-512747-23-00 (EU CTIS Number)
Record Dates: First submitted 2021-02-18; First posted 2021-02-25 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Transfusion-dependent Alpha-Thalassemia; Transfusion-dependent Beta-Thalassemia
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mitapivat (Experimental): Participants randomized to receive mitapivat 100 milligrams (mg), orally, twice daily (BID) for 48 weeks in the double-blind (DB) period and for up to 5 years in the open label extension (OLE) period.
  Interventions: Drug: Mitapivat
- Placebo (Placebo Comparator): Participants randomized to receive placebo matching mitapivat, orally, BID for 48 weeks in the DB period followed by mitapivat 100 mg, orally, BID for up to 5 years in the OLE period.
  Interventions: Drug: Placebo Matching Mitapivat; Drug: Mitapivat

INTERVENTIONS:
Drug: Placebo Matching Mitapivat — Tablets
  Arms: Placebo
Drug: Mitapivat — Tablets
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate

SUMMARY:
The primary objective of this study was to compare the effect of mitapivat versus placebo on transfusion burden in participants with α- or β-transfusion-dependent thalassemia.

DETAILED DESCRIPTION:
The mitapivat group included 171 participants. The placebo group included 87 participants.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to (≥)18 years of age at the time of providing informed consent;
* Documented diagnosis of thalassemia (β-thalassemia with or without α-globin gene mutations, hemoglobin E (HbE)/β-thalassemia, or α-thalassemia/hemoglobin H (HbH) disease) based on deoxyribonucleic acid (DNA) analysis;
* Considered transfusion-dependent, defined as 6 to 20 red blood cells (RBC) units transfused and ≤6-week transfusion-free period during the 24-week period before randomization;
* If taking hydroxyurea, the hydroxyurea dose must be stable for ≥16 weeks before randomization;
* Women of childbearing potential (WOCBP) must be abstinent of sexual activities that may induce pregnancy as part of their usual lifestyle or agree to use two forms of contraception, one of which must be considered highly effective, from the time of providing informed consent, throughout the study, and for 28 days after the last dose of study drug. The second form of contraception can be an acceptable barrier method;
* Written informed consent before any study-related procedures are conducted and willing to comply with all study procedures for the duration of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or parturient;
* Documented history of homozygous or heterozygous sickle hemoglobin (Hb S) or hemoglobin C (Hb C);
* Prior exposure to gene therapy or prior bone marrow or stem cell transplantation;
* Currently receiving treatment with luspatercept; the last dose must have been administered ≥36 weeks before randomization;
* Currently receiving treatment with hematopoietic stimulating agents; the last dose must have been administered ≥36 weeks before randomization;
* History of malignancy (active or treated) ≤5 years before providing informed consent, except for nonmelanomatous skin cancer in situ, cervical carcinoma in situ, or breast carcinoma in situ;
* History of active and/or uncontrolled cardiac or pulmonary disease ≤6 months before providing informed consent;
* Hepatobiliary disorders;
* Estimated glomerular filtration rate <45 milliliters per minute (mL/min)/1.73 meter (m)^2 by Chronic Kidney Disease Epidemiology Collaboration creatinine equation;
* Nonfasting triglycerides >440 milligrams per deciliter (mg/dL) (5 millimoles per liter [mmol/L]);
* Active infection requiring systemic antimicrobial therapy at the time of providing informed consent;
* Positive test for hepatitis C virus antibody (HCVAb) with evidence of active HCV infection, or positive test for hepatitis B surface antigen (HBsAg);
* Positive test for human immunodeficiency virus (HIV)-1 antibody (Ab) or HIV-2 Ab;
* History of major surgery (including splenectomy) ≤6 months before providing informed consent and/or a major surgical procedure planned during the study;
* Current enrollment or past participation (≤12 weeks before administration of the first dose of study drug or a timeframe equivalent to 5 half-lives of the investigational study drug, whichever is longer) in any other clinical study involving an investigational treatment or device;
* Receiving strong CYP3A4/5 inhibitors that have not been stopped for ≥5 days or a timeframe equivalent to 5 half-lives (whichever is longer); or strong CYP3A4 inducers that have not been stopped for ≥4 weeks or a timeframe equivalent to 5 half-lives (whichever is longer), before randomization;
* Receiving anabolic steroids that have not been stopped for at least 4 weeks before randomization. Testosterone replacement therapy to treat hypogonadism is allowed. The testosterone dose and preparation must be stable for ≥12 weeks before randomization;
* Known allergy, or other contraindication, to mitapivat or its excipients (microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, mannitol, and magnesium stearate, Opadry® II Blue [hypromellose, titanium dioxide, lactose monohydrate, triacetin, and Federal Food, Drug, and Cosmetic (FD&C) Blue #2]);
* Any medical, hematological, psychological, or behavioral condition(s) or prior or current therapy that, in the opinion of the Investigator, may confer an unacceptable risk to participating in the study and/or could confound the interpretation of the study data. Also excluded are:

  * Participants who are institutionalized by regulatory or court order
  * Participants with any condition(s) that could create undue influence (including but not limited to incarceration, involuntary psychiatric confinement, and financial or familial affiliation with the Investigator or Sponsor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2029-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (75):
- United States (10):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - San Diego Hospital, UC San Diego Health, La Jolla, California
  - Children's Hospital Oakland, Oakland, California
  - Stanford Medicine, Palo Alto, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Weill Cornell Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Penn Medicine - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Seattle Cancer Care Alliance, University of Washington, Seattle, Washington
- Brazil (2):
  - Hospital Das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto
  - GSH Banco de Sangue de São Paulo, São Paulo
- Bulgaria (5):
  - MHAT "Dr. Nikola Vasiliev" AD, Kyustendil
  - UMHAT "Dr. Georgi Stranski" Pleven, Pleven
  - UMHAT "Sveti Georgi" EAD, Plovdiv
  - SHATHD Sofia, Sofia
  - UMHAT "Prof. Dr. Stoyan Kirkovich", Stara Zagora
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Toronto General Hospital, University Health Network, Toronto, Ontario
- Rigshospitalet, Hovedstaden, Denmark
- France (4):
  - CHU Hôpital Henri Mondor, Créteil
  - Hôpital Edouard Herriot, CHU de Lyon, Lyon
  - CHU Hôpital de la Timone, Marseille
  - Hôpital Necker Enfants Malades, Paris
- Germany (3):
  - Charité - UB - CVK - Medizinische Klinik, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Leipzig, Leipzig
- Greece (5):
  - University General Hospital of Patras, Achaia
  - Laiko General Hospital, Athens
  - Children's Hospital Agia Sophia, National and Kapodistrian University of Athens Medical School, Athens
  - University Hospital of Ioannina, Ioannina
  - Ippokrateio General Hospital, Thessaloniki
- Italy (8):
  - Ospedale "A. Perrino" - Brindisi, Brindisi
  - Ospedale Pediatrico Microcitemico, Cagliari
  - Ospedale Sant'Anna, Ferrara
  - Ente Ospedaliero Ospedali Galliera, Genova
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - A.O.U Di Modena, Modena
  - AOU L. Vanvitelli Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - A.O.U. San Luigi Gonzaga, Orbassano
- Chronic Care Center, Beirut, Lebanon
- Malaysia (8):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Sultanah Aminah Johor Bahru, Johor Bahru
  - Hospital Queen Elizabeth, Kota Kinabalu, Kota Kinabalu
  - Hospital Tunku Azizah, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Hospital Ampang, Pandan Indah
  - Hospital Pulau Pinang, Pulau Pinang
- Netherlands (3):
  - Amsterdam Universitair Medisch Centrum, Locatie AMC, Amsterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Erasmus MC, Westzeedijk 353
- Saudi Arabia (2):
  - King Abdullah International Medical Research Center, Riyadh
  - King Khalid University Hospital, Riyadh
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
- National Taiwan University Hospital, Taipei, Taiwan
- Thailand (7):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Faculty of Medicine Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Naresuan University Hospital, Mueang Phitsanulok
  - King Chulalongkorn Memorial Hospital, Pathum Wan
- Turkey (Türkiye) (6):
  - Acibadem Adana Hospital, Adana
  - Akdeniz University Faculty of Medicine, Antalya
  - Çukurova University, Balcalı
  - Ege University Faculty of Medicine, Bornova
  - Istanbul University Faculty of Medicine, Fatih
  - Hacettepe University, Mersin
- Burjeel Medical City, Abu Dhabi, United Arab Emirates
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 81 study sites in Malaysia,Taiwan,Thailand,Bulgaria,Brazil,Lebanon,Saudi Arabia,Turkey,United Arab Emirates,Canada, the United States,Denmark,France,Germany,Greece,Italy,Netherlands,Spain and the United Kingdom.Results are reported for 48-week DB period until primary completion date.Analysis of data for OLE period is still ongoing with anticipated completion in June 2029.Results for OLE period will be reported by June 2030.
Pre-assignment Details: A total of 305 participants with a diagnosis of Transfusion-Dependent Alpha- or Beta-Thalassemia (α- or β-TDT) were screened. Of which, 258 were randomized and 257 received study treatment in this study.
Groups:
- Mitapivat: Participants randomized to receive mitapivat 100 milligrams (mg), orally, twice daily (BID) for 48 weeks in double-blind period.
- Placebo: Participants randomized to receive placebo matching mitapivat, orally, BID for 48 weeks in double-blind period.
Period: Overall Study
Arm/Group | Mitapivat | Placebo
Started | 171 | 87
Safety Analysis Set (Safety Analysis Set: all participants who received at least 1 dose of study treatment. If a participant randomized to placebo received at least 1 dose of mitapivat in the double-blind period, then the participant is classified to the mitapivat arm. One participant, randomized to placebo, received mitapivat and was classified in the mitapivat arm in the safety analysis set.) | 172 | 85
Completed | 155 | 83
Not Completed | 16 | 4
Not completed — Randomized, never treated | 0 | 1
Not completed — Adverse Event | 9 | 1
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Mitapivat: Participants randomized to receive mitapivat 100 mg, orally, BID for 48 weeks in double-blind period.
- Total: Total of all reporting groups
Arm/Group | Mitapivat | Placebo | Total
Number analyzed (Participants) | 171 | 87 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (11.61) | 34.7 (9.77) | 35.5 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 43 | 136
  Male | 78 | 44 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 158 | 79 | 237
  Unknown or Not Reported | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 99 | 56 | 155
  Asian | 56 | 22 | 78
  Black or African American | 1 | 1 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Multiracial | 2 | 0 | 2
  Unknown | 7 | 3 | 10
  Not reported | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Double-blind Period: Percentage of Participants Who Achieved Transfusion Reduction Response (TRR)
Description: TRR is defined as ≥50% reduction in transfused red blood cells (RBC) units with a reduction of ≥2 units of transfused RBCs in any consecutive 12-week period through Week 48 compared with baseline transfusion burden standardized to 12 weeks. Baseline transfusion burden standardized to 12 weeks= (12/24) × total number of RBC units transfused during 24-week period before the randomization date for participants randomized and not dosed or the start of study treatment for participants randomized and dosed. Participants withdrawn from the study before Week 12 (Day 85) were considered nonresponders.
Time Frame: Double-blind Period: Baseline through Week 48
Population: FAS included all participants who were randomized.
Measure: Number; unit: percentage of participants
Groups:
- Mitapivat: Participants randomized to receive mitapivat 100 mg, orally, BID for 48 weeks in the double-blind period.
- Placebo: Participants randomized to receive placebo matching mitapivat, orally, BID for 48 weeks in the double-blind period.
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 171 | 87
percentage of participants | 30.4 | 12.6
Statistical Analysis 1: Comparison: Mitapivat vs Placebo; The p-value is based on the Mantel-Haenszel stratum weighted method adjusting for randomization stratification factors; Test type: Superiority; p = 0.0003, Mantel Haenszel; Common Risk Difference on Response Rate = 17.6, 95% CI 2-sided [8.0 to 27.2]

2. Secondary Outcome: Double-blind Period: Percentage of Participants Who Achieved TRR2
Description: TRR2, defined as a ≥50% reduction in transfused RBC units in any consecutive 24-week period through Week 48 compared with the 24-week baseline transfusion burden, is reported. Baseline transfusion burden standardized to 24 weeks is the total number of RBC units transfused during the 24-week period before the randomization date for participants randomized and not dosed or the start of study treatment for participants randomized and dosed. Participants withdrawn from the study before Week 24 (Day 169) were considered nonresponders.
Time Frame: Double-blind period: Baseline through Week 48
Population: FAS included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 171 | 87
percentage of participants | 13.5 | 2.3
Statistical Analysis 1: Comparison: Mitapivat vs Placebo; The p-value is based on the Mantel-Haenszel stratum weighted method adjusting for randomization stratification factors; Test type: Superiority; p = 0.0003, Mantel Haenszel; Common Risk Difference on Response Rate = 11.1, 95% CI 2-sided [5.1 to 17.0]

3. Secondary Outcome: Double-blind Period: Percentage of Participants Who Achieved TRR3
Description: TRR3, defined as a ≥33% reduction in transfused RBC units from Week 13 through Week 48 compared with the baseline transfusion burden standardized to 36 weeks, is reported. Baseline transfusion burden standardized to 36 weeks= (36/24) × total number of RBC units transfused during the 24-week period before the randomization date for participants randomized and not dosed or the start of study treatment for participants randomized and dosed. Participants withdrawn from the study before Week 48 were considered nonresponders.
Time Frame: Double-blind period: Baseline up to Week 13 through Week 48
Population: FAS included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 171 | 87
percentage of participants | 14.6 | 1.1
Statistical Analysis 1: Comparison: Mitapivat vs Placebo; The p-value is based on the Mantel-Haenszel stratum weighted method adjusting for randomization stratification factors; Test type: Superiority; p < 0.0001, Mantel Haenszel; Common Risk Difference on Response Rate = 13.4, 95% CI 2-sided [7.7 to 19.1]

4. Secondary Outcome: Double-blind Period: Percentage of Participants Who Achieved TRR4
Description: TRR4, defined as a ≥50% reduction in transfused RBC units from Week 13 through Week 48 compared with the baseline transfusion burden standardized to 36 weeks, is reported. Baseline transfusion burden standardized to 36 weeks = (36/24) × total number of RBC units transfused during the 24-week period before the randomization date for participants randomized and not dosed or the start of study treatment for participants randomized and dosed. Participants withdrawn from the study before Week 48 were considered nonresponders.
Time Frame: Double-blind period: Baseline up to Week 13 through Week 48
Population: FAS included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 171 | 87
percentage of participants | 7.6 | 1.1
Statistical Analysis 1: Comparison: Mitapivat vs Placebo; The p-value is based on the Mantel-Haenszel stratum weighted method adjusting for randomization stratification factors; Test type: Superiority; p = 0.0056, Mantel Haenszel; Common Risk Difference on Response Rate = 6.4, 95% CI 2-sided [1.9 to 10.9]

5. Secondary Outcome: Double-blind Period: Percent Change From Baseline in Transfused RBC Units
Description: Transfusion burden from Week 13 through Week 48 standardized to 36 weeks is defined as number of transfused RBC units from Day 85 through Week 48 in the Double-blind Period ×36/(Number of days from Day 85 through Week 48 in the Double-blind Period/7). Baseline transfusion burden standardized to 36 weeks= (36/24)× is the total number of RBC units transfused during the 24-week period before the randomization date for participants randomized and not dosed or within 168 days before the start of study treatment for participants randomized and dosed.
Time Frame: Double-blind Period: Baseline, Week 13 through Week 48
Population: FAS included all participants who were randomized. Overall number of participants analyzed indicates number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 155 | 83
percent change | 10.96 (2.149) | 3.32 (2.846)

6. Secondary Outcome: Double-blind Period: Percentage of Participants Who Achieved Transfusion-Independence
Description: Transfusion-independence is defined as transfusion-free for ≥8 consecutive weeks through Week 48 in the double-blind period.
Time Frame: Double-blind Period: Baseline through Week 48
Population: FAS included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 171 | 87
percentage of participants | 9.9 | 1.1

7. Secondary Outcome: Double-blind Period: Change From Baseline in Iron Levels
Description: Iron metabolism was assessed based on Iron levels.
Time Frame: Double-blind Period: Baseline through Week 48
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: micromoles per liter (µmol/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 149 | 75
micromoles per liter (µmol/L) | -4.57 (0.949) | 2.06 (1.280)

8. Secondary Outcome: Double-blind Period: Change From Baseline in Serum Ferritin Levels
Description: Iron metabolism was assessed based on serum ferritin levels.
Time Frame: Double-blind Period: Baseline through Week 48
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: micrograms per liter (µg/L)
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 148 | 75
micrograms per liter (µg/L) | 45.3 (88.90) | 76.3 (119.84)

9. Secondary Outcome: Double-blind Period: Change From Baseline in Total Iron Binding Capacity
Description: Iron metabolism was assessed based on total iron binding capacity.
Time Frame: Double-blind Period: Baseline through Week 48
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: µmol/L
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 80 | 41
µmol/L | -21.80 (3.597) | -1.23 (5.053)

10. Secondary Outcome: Double-blind Period: Change From Baseline in Transferrin Saturation (TSAT) Levels
Description: Iron metabolism was assessed based on TSAT levels. Transferrin saturation is reported by dividing value of serum iron by total iron binding capacity.
Time Frame: Double-blind Period: Baseline through Week 48
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 80 | 40
Ratio | 0.079 (0.0261) | -0.013 (0.0371)

11. Secondary Outcome: Double-blind Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Related TEAEs and TEAEs With Severity Greater Than or Equal to Grade 3
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study drug. A serious adverse event (SAE) is any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are AEs with an initial onset date during the on-treatment period or worsening from baseline and includes both serious & non-serious TEAEs. Severity of AEs was evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03): grade 1: mild; grade 2: moderate; grade 3: severe or medically significant but not immediately life-threatening; grade 4: life threatening or disabling; grade 5: death related to AE.
Time Frame: Double-blind Period: From first dose of study drug up to week 48
Population: Safety Analysis Set (SAS) included all participants who had received at least 1 dose of study treatment. Participants were classified according to the treatment received. If a participant was randomized to placebo and received at least 1 dose of mitapivat in the double-blind period, then the participant was classified to the mitapivat arm. One subject, randomized to placebo, received mitapivat and was classified in the mitapivat arm in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 172 | 85
Participants
  Participants with TEAEs | 155 | 71
  Participants with serious TEAEs | 19 | 13
  Participants with TEAEs related to study drug | 65 | 16
  Participants with any TEAE of Grade ≥ 3 | 32 | 12

12. Secondary Outcome: Open-label Extension Period: Number of Participants With TEAEs, Serious TEAEs, Related TEAEs, Related TEAEs and TEAEs With Severity of Greater Than or Equal to 3
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with the study drug. A serious adverse event (SAE) is any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are AEs with an initial onset date during the on-treatment period or worsening from baseline and includes both serious & non-serious TEAEs. Severity of abnormalities was evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE; Version 4.03): grade 1: mild; grade 2: moderate; grade 3: severe or medically significant but not immediately life-threatening; grade 4: life threatening or disabling; grade 5: death related to AE.
Time Frame: Open-Label Extension Period: From Week 48 up to end of study (approximately 5 years)
Reporting Status: Not Posted, anticipated posting 2030-06

13. Secondary Outcome: Double-blind Period: Plasma Concentrations of Mitapivat
Time Frame: Double-blind Period: Pre-dose at Week 12; pre-dose at Week 24; pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 36
Population: Pharmacokinetic (PK) Analysis Set included a subset of the safety analysis set and included all participants with at least 1 mitapivat plasma concentration measurement ≥ lower limit of quantification (LLQ). Number analyzed signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Mitapivat
Number analyzed (Participants) | 165
nanograms per milliliter (ng/mL)
  Pre-dose at Week 12: number analyzed (Participants) | 142
  Pre-dose at Week 12 | 122.90 (252.666)
  Pre-dose at Week 24: number analyzed (Participants) | 143
  Pre-dose at Week 24 | 96.55 (184.835)
  Pre-dose at Week 36: number analyzed (Participants) | 153
  Pre-dose at Week 36 | 129.31 (260.610)
  0.5 Hour Post-dose at Week 36: number analyzed (Participants) | 150
  0.5 Hour Post-dose at Week 36 | 1282.21 (1007.068)
  1 Hour Post-dose at Week 36: number analyzed (Participants) | 147
  1 Hour Post-dose at Week 36 | 1468.69 (713.248)
  3 Hours Post-dose at Week 36: number analyzed (Participants) | 149
  3 Hours Post-dose at Week 36 | 765.32 (372.719)
  5 Hours Post-dose at Week 36: number analyzed (Participants) | 148
  5 Hours Post-dose at Week 36 | 371.11 (232.556)
  7 Hours Post-dose at Week 36: number analyzed (Participants) | 143
  7 Hours Post-dose at Week 36 | 221.78 (172.845)

14. Secondary Outcome: Double-blind Period: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-last) of Mitapivat
Description: Area under the concentration-time curve from time zero to Tlast on dosing day, calculated using the linear-log trapezoidal rule.
Time Frame: Double-blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 36
Population: PK analysis set is a subset of the safety analysis set and included all participants with at least 1 plasma mitapivat concentration measurement ≥LLQ. Overall number of participants analyzed indicates number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Mitapivat
Number analyzed (Participants) | 141
hours*nanograms per milliliter (h*ng/mL) | 4365.84 (35.9)

15. Secondary Outcome: Double-blind Period: Maximum Observed Plasma Concentration (Cmax) of Mitapivat
Time Frame: Double-blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose Week 36
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Mitapivat
Number analyzed (Participants) | 149
nanograms per milliliter (ng/mL) | 1603.00 (45.6)

16. Secondary Outcome: Double-blind Period: Time to Reach of Maximum Observed Plasma Concentration (Tmax) of Mitapivat
Time Frame: Double-blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose Week 36
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Mitapivat
Number analyzed (Participants) | 149
Hours | 1.000 [0.42 to 5.00]

17. Secondary Outcome: Double-blind Period: Time of Last Quantifiable Concentration (Tlast) of Mitapivat
Time Frame: Double-blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose Week 36
Population: as for outcome 14
Measure: Median (Full Range); unit: Hours
Arm/Group | Mitapivat
Number analyzed (Participants) | 147
Hours | 6.750 [4.83 to 7.17]

18. Secondary Outcome: Double-blind Period: Last Quantifiable Plasma Concentration (Clast) of Mitapivat
Description: Clast is the last quantifiable concentration after a single dose or within the dosing interval (tau) for multiple doses.
Time Frame: Double-blind Period: Pre-dose, 0.5, 1, 3, 5, 7 hours post-dose Week 36
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mitapivat
Number analyzed (Participants) | 147
ng/mL | 175.76 (85.1)

19. Secondary Outcome: Double-blind Period: Blood Concentration of Adenosine Triphosphate (ATP)
Time Frame: Double-blind Period: Pre-dose at Day 1; pre-dose at Week 12; pre-dose at Week 24; pre-dose, 0.5, 1, 3, 5, 7 hours post-dose at Week 36
Population: Pharmacodynamic (PD) analysis set is a subset of the safety analysis set and included all participants with at least 1 blood 2,3-diphosphoglycerate (DPG) or ATP concentration measurement ≥ LLQ. Number analyzed signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 169 | 85
µg/mL
  Pre-dose at Day 1: number analyzed (Participants) | 123 | 64
  Pre-dose at Day 1 | 224.33 (40.031) | 236.23 (47.368)
  Pre-dose at Week 12: number analyzed (Participants) | 135 | 64
  Pre-dose at Week 12 | 283.39 (59.217) | 204.19 (33.207)
  Pre-dose at Week 24: number analyzed (Participants) | 136 | 74
  Pre-dose at Week 24 | 279.16 (53.652) | 200.84 (30.333)
  Pre-dose at Week 36: number analyzed (Participants) | 148 | 73
  Pre-dose at Week 36 | 280.72 (61.834) | 210.47 (43.330)
  0.5 Hour Post-dose at Week 36: number analyzed (Participants) | 144 | 65
  0.5 Hour Post-dose at Week 36 | 274.75 (63.513) | 206.83 (39.389)
  1 Hour Post-dose at Week 36: number analyzed (Participants) | 141 | 66
  1 Hour Post-dose at Week 36 | 277.45 (58.668) | 209.92 (38.597)
  3 Hours Post-dose at Week 36: number analyzed (Participants) | 143 | 67
  3 Hours Post-dose at Week 36 | 281.70 (61.262) | 213.63 (43.949)
  5 Hours Post-dose at Week 36: number analyzed (Participants) | 142 | 68
  5 Hours Post-dose at Week 36 | 283.76 (61.216) | 208.18 (40.965)
  7 Hours Post-dose at Week 36: number analyzed (Participants) | 140 | 60
  7 Hours Post-dose at Week 36 | 281.47 (57.163) | 212.02 (45.767)

20. Secondary Outcome: Double-blind Period: Blood Concentration of 2,3 - Diphosphoglycerate (2,3-DPG)
Time Frame: as for outcome 19
Population: PD analysis set is a subset of the safety analysis set and included all participants with at least 1 blood 2,3-diphosphoglycerate (2,3-DPG) or adenosine triphosphate (ATP) concentration measurement ≥LLQ. Number analyzed signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Mitapivat | Placebo
Number analyzed (Participants) | 169 | 85
µg/mL
  Pre-dose at Day 1: number analyzed (Participants) | 123 | 64
  Pre-dose at Day 1 | 426.67 (75.055) | 417.13 (87.448)
  Pre-dose at Week 12: number analyzed (Participants) | 134 | 65
  Pre-dose at Week 12 | 274.25 (76.114) | 365.88 (67.238)
  Pre-dose at Week 24: number analyzed (Participants) | 136 | 75
  Pre-dose at Week 24 | 275.60 (78.307) | 355.57 (59.420)
  Pre-dose at Week 36: number analyzed (Participants) | 148 | 73
  Pre-dose at Week 36 | 289.11 (78.658) | 368.81 (71.481)
  0.5 Hour Post-dose at Week 36: number analyzed (Participants) | 145 | 65
  0.5 Hour Post-dose at Week 36 | 286.06 (73.409) | 367.74 (62.673)
  1 Hour Post-dose at Week 36: number analyzed (Participants) | 142 | 67
  1 Hour Post-dose at Week 36 | 281.73 (80.276) | 368.67 (66.037)
  3 Hours Post-dose at Week 36: number analyzed (Participants) | 144 | 67
  3 Hours Post-dose at Week 36 | 280.93 (76.916) | 383.00 (91.727)
  5 Hours Post-dose at Week 36: number analyzed (Participants) | 142 | 68
  5 Hours Post-dose at Week 36 | 272.73 (65.327) | 359.09 (72.144)
  7 Hours Post-dose at Week 36: number analyzed (Participants) | 139 | 62
  7 Hours Post-dose at Week 36 | 268.17 (65.942) | 369.19 (75.546)

ADVERSE EVENTS:
Time Frame: Double-blind period: From first dose of study drug up to week 48
Description: AEs: Safety Analysis Set (SAS) was used. One participant, randomized to placebo, received mitapivat and is classified in the mitapivat arm in the SAS. All-Cause Mortality: FAS was used. Safety data are presented for Double-blind Period only. The OLE period is ongoing with anticipated completion in June 2029. Results for OLE will be reported separately by June 2030.
Arm/Group | Mitapivat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/87
Serious Adverse Events (participants affected / at risk) | 19/172 | 13/85
Other Adverse Events (participants affected / at risk) | 122/172 | 50/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitapivat (N=172) | Placebo (N=85)
Pneumonia (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 0 | 1
Splenic haematoma (Blood and lymphatic system disorders) | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 1 | 0
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Limb deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mitapivat (N=172) | Placebo (N=85)
Upper respiratory tract infection (Infections and infestations) | 27 | 14
Influenza (Infections and infestations) | 14 | 4
Nasopharyngitis (Infections and infestations) | 11 | 4
Urinary tract infection (Infections and infestations) | 11 | 0
COVID-19 (Infections and infestations) | 8 | 8
Headache (Nervous system disorders) | 46 | 10
Fatigue (General disorders) | 18 | 2
Pyrexia (General disorders) | 17 | 6
Asthenia (General disorders) | 10 | 4
Influenza like illness (General disorders) | 9 | 2
Diarrhoea (Gastrointestinal disorders) | 19 | 7
Nausea (Gastrointestinal disorders) | 13 | 5
Vomiting (Gastrointestinal disorders) | 8 | 7
Initial insomnia (Psychiatric disorders) | 24 | 4
Middle insomnia (Psychiatric disorders) | 10 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT04770779/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT04770779/SAP_001.pdf